CLINICAL TRIAL: NCT04704271
Title: Gender Related Differences in the Acute Effects of Delta-9-Tetrahydrocannabinol in Healthy Humans: Sub-Study II
Acronym: THC-Gender-II
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1505015940.B
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delta-9-Tetrahydrocannabinol (THC) (Active Comparator): 4 mg vaporized THC will be administered.
  Interventions: Drug: Inhaled THC
- Placebo (Placebo Comparator): Inhaled placebo (no active cannabinoids)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled THC — 4 mg inhaled THC
  Other Names: Delta-9-Tetrahydrocannabinol
  Arms: Delta-9-Tetrahydrocannabinol (THC)
Drug: Placebo — Inhaled placebo (no active cannabinoids)
  Arms: Placebo

SUMMARY:
The purpose of the study is to characterize the acute effects of cannabinoids in women relative to men and to begin probing the mechanisms that may underlie gender differences.

DETAILED DESCRIPTION:
To characterize the acute effects of vaporized THC in women relative to men and to begin probing the mechanisms that may underlie gender differences.

ELIGIBILITY:
Inclusion Criteria:

* At least one lifetime exposure to cannabis
* Good physical and mental health

Exclusion Criteria:

* Cannabis naïve individuals
* Major current or recent stressors

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline: Rewarding Effects measured by Visual Analog Scale (VAS) | Changes in "high" assessed over the following timepoints: baseline, +60, +80, +120, +180, +300 minutes after start of oral Dronabinol administration.
  Subjective measure of THC induced "high"
Change from Baseline: Verbal Learning: Measured by Rey Auditory Verbal Learning Test (RAVLT) | Baseline and +80 minutes after start of oral Dronabinol administration.
  Measured as delay recall on the AVLT

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit at the VA Connecticut Healthcare System, Yale School of Medicine, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No